CLINICAL TRIAL: NCT06144242
Title: Randomized-controlled Trial to Assess Whether Feedback on a New Stewardship Metric Can Improve Antibiotic-prescribing for Acute Respiratory Tract Infections in Urgent Care Clinics
Brief Title: Improving Antibiotic Use for ARIs in Urgent Care Clinics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Livorsi (Other)
Responsible Party: Sponsor-Investigator, Daniel Livorsi, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202308456
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Antibacterial Agents; Ambulatory Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback on RTD metric (Experimental): An e-mail will be sent to the clinicians in the experimental arm every two months describing their performance on the RTD metric and making a comparison to how their peers have performed. The e-mail will also direct clinicians to visit a dashboard to review their practice in greater depth.
  Interventions: Behavioral: Feedback on RTD metric
- No feedback on RTD metric (No Intervention): Any clinician assigned to the control arm will not receive the above-mentioned e-mails.

INTERVENTIONS:
Behavioral: Feedback on RTD metric — Clinicians in the experimental arm will receive feedback on the RTD metric while clinicians in the No intervention arm will not.
  Arms: Feedback on RTD metric

SUMMARY:
Many clinicians prescribe antibiotics for patients with acute respiratory infections even when antibiotics will not benefit the patient because the infection is due to a virus. To discourage this type of unnecessary antibiotic use, the investigators will assess whether it is helpful to give clinicians feedback on how often they prescribe antibiotics for respiratory infections in comparison to their peers. The investigators will perform this study across Urgent Care and QuickCare clinics within a single healthcare system.

DETAILED DESCRIPTION:
The investigators have used an established HEDIS (Healthcare Effectiveness Data and Information Set) metric to evaluate Urgent Care and QuickCare clinicians on their antibiotic use for respiratory tract diagnoses (RTDs). This RTD metric excludes visits that are more complicated, based on well-defined criteria. Based on our baseline assessment (2018-2022), the investigators estimate that most clinicians in this setting are frequently prescribing unnecessary antibiotics.

The investigators will perform a randomized controlled trial to assess whether providing individualized feedback to clinicians on the RTD metric can safely reduce antibiotic use for qualifying respiratory tract visits across Urgent and QuickCare settings within a single integrated healthcare system. Clinicians who do not opt-out of the trial will be randomized to either receive feedback or not receive feedback on this RTD metric. The trial will last for 18 months. The primary outcome of effectiveness will be the frequency of antibiotic-prescribing for RTD visits. Secondary outcomes include total antibiotic use (regardless of diagnosis), changes in the use of diagnostic codes, 30-day rates of follow-up visits and hospital admissions. The RE-AIM framework will be used to guide additional study evaluation.

ELIGIBILITY:
Any clinician who works in Urgent Care or QuickCare clinics within our healthcare system.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of antibiotic-prescribing for RTD visits | 24 hours of visit
  Percentage of all qualifying respiratory tract diagnosis (RTD) visits prescribed an antibiotic

SECONDARY OUTCOMES:
Frequency of antibiotic-prescribing for all visits | 24 hours of visit
  Percentage of all visits prescribed an antibiotic, regardless of the diagnosis
Follow-up visit to Urgent Care or QuickCare | 30 days
  Percentage of patients with a qualifying RTD visit who were seen at least once in Urgent Care or QuickCare within the 30 days after their index visit date.
Follow-up Emergency Department visit and/or acute-care hospitalization | 30 days
  Percentage of patients with a qualifying RTD visit who were seen at least once in the Emergency Department and/or who were hospitalized (any reason) within the 30 days after their index visit date.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT06144242/Prot_SAP_000.pdf